CLINICAL TRIAL: NCT02779452
Title: Does Brain Functions Depend on Omega 3 Transferred to the Fetus During the Intra Uterine Life ?
Brief Title: Gestational Diabetes Mellitus and Neurodevelopment in Newborns
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, PhD, Université de Sherbrooke
Other Study IDs: GDM and neurodevelopment
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes, Gestational; Glucose Metabolism Disorders
Keywords: neurodevelopment; electroencephalography; gestational diabetes mellitus; omega 3 polyunsaturated fatty acids
MeSH Terms: conditions — Diabetes, Gestational; Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cord blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GDM newborns: Newborns from gestational diabetes mellitus pregnancy
- No GDM newborns: Newborn from a normal pregnancy

SUMMARY:
The purpose of this study is to evaluate the feasibility of using a quantitative EEG method to evaluate neurodevelopment in newborns and to evaluate whether subtle neurodevelopmental deficits can be detected in newborns from mothers with gestational diabetes mellitus (GDM) compared to control newborns.

The second purpose of this study is to determine whether cord blood concentration in docosahexaenoic acid (DHA), an omega-3 fatty acid, is similar in neonates of well-controlled mothers with gestational diabetes mellitus (GDM) compared to control mothers, and to evaluate whether this contributes to neonates neurodevelopment status.

DETAILED DESCRIPTION:
Maternal weight is measured close to delivery and BMI is calculated. Birth weight, length, head circumference, Apgar score and glycaemia are recorded at birth. An EEG are performed on the newborn within 48 hrs after birth.A maternal blood sample is collected at admission to measure maternal glycated hemoglobin (A1C). Cord blood samples are collected in the umbilical vein after delivery.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* aged between 18 and 40 years

Exclusion Criteria:

* smoking,
* illicit drug consumption,
* omega-3/6 consumption,
* liver or renal disease,
* cancer
* any medical conditions affecting glucose/lipid metabolism.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with singleton pregnancy were recruited in the Centre Hospitalier Universitaire de Sherbrooke (CHUS) at 24 - 28 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in neurodevelopment | At birth
  Evaluate change in neurodevelopment with GDM

SECONDARY OUTCOMES:
Change in DHA level in cord blood | At birth
  Evaluate change in DHA level with GDM

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Plourde, PhD, Principal Investigator — Université de Sherbrooke

IPD SHARING:
Plan to Share IPD: No